CLINICAL TRIAL: NCT04272567
Title: Norepinephrine Prophylaxis for Postspinal Anesthesia Hypotension in Parturients Undergoing Cesarean Section: a Randomized, Placebo-controlled Dose-finding Trial
Brief Title: Norepinephrine Prophylaxis for Postspinal Anesthesia Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Yi Chen-2020-1
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-02

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Hypotension; Cesarean section; Dose-finding
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Vasoconstrictor Agents; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Sham Comparator): Simultaneous with subarachnoid block, a bolus of 1ml normal saline was given followed by normal saline infusion
  Interventions: Drug: Normal saline
- 0.025 μg/kg/min group (Experimental): Simultaneous with subarachnoid block, a bolus of 6μg norepinephrine was given followed by a maintenance dose of norepinephrine (0.025 μg/kg/min).
  Interventions: Drug: Norepinephrine
- 0.05 μg/kg/min group (Experimental): Simultaneous with subarachnoid block, a bolus of 6μg norepinephrine was given followed by a maintenance dose of norepinephrine (0.05 μg/kg/min).
  Interventions: Drug: Norepinephrine
- 0.075 μg/kg/min group (Experimental): Simultaneous with subarachnoid block, a bolus of 6μg norepinephrine was given followed by a maintenance dose of norepinephrine (0.075 μg/kg/min).
  Interventions: Drug: Norepinephrine
- 0.1 μg/kg/min group (Experimental): Simultaneous with subarachnoid block, a bolus of 6μg norepinephrine was given followed by a maintenance dose of norepinephrine (0.1 μg/kg/min).
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Simultaneous with subarachnoid block, a bolus of 6μg norepinephrine was given followed by different infusion dose of norepinephrine.
  Other Names: Vasopressors
  Arms: 0.025 μg/kg/min group; 0.05 μg/kg/min group; 0.075 μg/kg/min group; 0.1 μg/kg/min group
Drug: Normal saline — Simultaneous with subarachnoid block, a bolus of 1ml normal saline was given followed by normal saline infusion
  Other Names: NS
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate the suitable infusion dose of norepinephrine for prophylaxis against post-spinal anesthesia hypotension.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Vasopressors has been highly recommended for routine prevention and/or treatment of post-spinal anesthesia hypotension. As a potential substitute drug for phenylephrine, norepinephrine has gradually been used in parturients undergoing cesarean section. There's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. But the ideal infusion dose of norepinephrine is still unknown. The purpose of this study is to investigate the suitable infusion dose of norepinephrine for prophylaxis against post-spinal anesthesia hypotension.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
Overall stability of systolic blood pressure control versus baseline | 1-15 minutes after spinal anesthesia.
  Evaluated by performance error (PE).
Overall stability of heart rate control versus baseline | 1-15 minutes after spinal anesthesia.
  Evaluated by performance error (PE).
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia.
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia.
  Heart rate < 55 beats/min.
The incidence of hypertension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery.
  From umbilical arterial blood gases.
Partial pressure of oxygen | Immediately after delivery.
  From umbilical arterial blood gases.
Base excess | Immediately after delivery.
  From umbilical arterial blood gases.
APGAR score | 1min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Dr., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China